CLINICAL TRIAL: NCT05749393
Title: Effect of Heparinization on Intracranial Aneurysm
Brief Title: Effect of Different Heparinization Schemes on Prognosis of Intracranial Aneurysm
Acronym: EODHS-IA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Lu Hua, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EODHS-IA
Record Dates: First submitted 2023-02-17; First posted 2023-03-01 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Intracranial Aneurysm
Keywords: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm | interventions — Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-dose group (Experimental): The initial dose was 50U/kg intravenous injection, and the dosage was halved by intravenous injection every 1 hour to the minimum 1000u/h. The medication will be discontinued at the end of the procedure.
  Interventions: Drug: Heparin sodium
- High-dose group (Experimental): The initial dose was 70U/kg intravenous injection, and the dosage was halved by intravenous injection every 1 hour to the minimum 1000u/h. The medication will be discontinued at the end of the procedure.
  Interventions: Drug: Heparin sodium

INTERVENTIONS:
Drug: Heparin sodium — Intravenous heparin was administered during intracranial aneurysm embolization with a guide catheter and discontinued at the end of the procedure.

SUMMARY:
The goal of this clinical trial is to compare intracranial aneurysm patients. The main question it aims to answer are: Which heparinization regimen is most beneficial to patients during surgery for intracranial aneurysms. Participants will be randomized to different intraoperative heparinization regimens: (i) 50 U/kg intravenous (IV) at 1-h intervals reduced by half to a minimum of 1000 u/h; (ii) 70 U/kg IV at 1-h intervals reduced by half to a minimum of 1000 u/h. MRI will be performed within 72 h after surgery, and the DWI sequence of MRI will be analyzed. If there is a comparison group: Researchers will compare different intraoperative heparinization protocol groups to see which dose of intraoperative heparin has the best prognosis for use.

ELIGIBILITY:
Inclusion Criteria:

1. Greater than 18 years old, less than 75 years old
2. Patients with unruptured intracranial aneurysm were confirmed by DSA.
3. Coagulation function should be normal in the enrolled patients.

Exclusion Criteria:

1. Dissection aneurysm, blister aneurysm, moyamoya disease or arteriovenous malformation.
2. Previous use of antithrombotic drugs (including anticoagulant or antiplatelet aggregation drugs).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-04-30 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Size of the ischemic focus | This will be evaluated within 24 hours after the procedure.
  Cranial MRI will be performed on postoperative patients within 24 hours. The presence of high signal on diffusion weighted imaging sequences indicated the occurrence of cerebral infarction.

CONTACTS AND LOCATIONS:
Overall Officials: Hua Lu, Doctor, Principal Investigator — First Affiliated Hospital, Nanjing Medical University
Locations (1):
- Jiangsu Province Hospital, Nanjing, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be available to other researchers under the approval of the ethical committee.
Supporting Information: Study Protocol, CSR
Time Frame: the data will be available when summary data are published.

REFERENCES:
- [Background] Zhang L, Zhou X, Liu Y, Ding C, Wang Y, Yang H. The Utility of Diffusion-Weighted MRI Lesions to Compare the Effects of Different Heparinization Schemes in Intracranial Aneurysms Treated by Endovascular Intervention. Front Neurol. 2020 Dec 10;11:609384. doi: 10.3389/fneur.2020.609384. eCollection 2020. PMID 33424758
- [Background] Narata AP, Amelot A, Bibi R, Herbreteau D, Angoulvant D, Gruel Y, Janot K. Dual Antiplatelet Therapy Combining Aspirin and Ticagrelor for Intracranial Stenting Procedures: A Retrospective Single Center Study of 154 Consecutive Patients With Unruptured Aneurysms. Neurosurgery. 2019 Jan 1;84(1):77-83. doi: 10.1093/neuros/nyy002. PMID 29490066